CLINICAL TRIAL: NCT05716945
Title: Optimized Immunosuppression for Corneal Transplantation: A Multi-center Randomized Controlled Clinical Trial
Brief Title: The OPTIMISE Study
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-500109-41-00
Record Dates: First submitted 2023-01-30; First posted 2023-02-08 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Pseudophakic Bullous Keratopathy; Fuchs' Endothelial Dystrophy; Intraocular Pressure
Keywords: Descemet Stripping Endothelial Keratoplasty; Cornea
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy; Corneal Diseases | interventions — Fluorometholone; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Intervention STEP I (Year 1 after DMEK) (Experimental)
  Interventions: Drug: Fluorometholone 0.1% Oph Susp; Drug: Dexamethasone 0.1% ophthalmic suspension
- Control STEP I (Year 1 after DMEK) (Active Comparator)
  Interventions: Drug: Dexamethasone 0.1% ophthalmic suspension
- Intervention STEP II (Year 2 after DMEK) (Experimental)
  Interventions: Other: Stop steroids
- Control STEP II (Year 2 after DMEK) (Active Comparator)
  Interventions: Drug: Fluorometholone 0.1% Oph Susp

INTERVENTIONS:
Drug: Fluorometholone 0.1% Oph Susp — Year 1: DMS 0.1% 6 times a day for 1 month followed by FML 0.1% 4 times a day for two months tapered off to once daily within four months and then once a day for 6 months.
  Year 2: Half the patients in each study arm will use FML 0.1% daily.
  Arms: Control STEP II (Year 2 after DMEK); Intervention STEP I (Year 1 after DMEK)
Drug: Dexamethasone 0.1% ophthalmic suspension — Year 1: DMS 0.1% 6 times a day for 1 month tapered off to once daily within 6 months and then once a day for 6 months.
  Arms: Control STEP I (Year 1 after DMEK); Intervention STEP I (Year 1 after DMEK)
Other: Stop steroids — Half the patients in each study arm will discontinue steroids.
  Arms: Intervention STEP II (Year 2 after DMEK)

SUMMARY:
Rationale:

The cornea is the most transplanted tissue in the Netherlands, with more than 1,500 procedures performed each year. A minimally invasive technique called Descemet Membrane Endothelial Keratoplasty (DMEK) has become the preferred method in the past decade. The main advantage of DMEK over previous techniques is a low graft rejection rate (1-2% per year). Despite this, rejection prophylaxis after DMEK follows the same high potency regimen as previous techniques in the first year, and patients are burdened with indefinite immunosuppression. The current project, OPTIMISE, aims to establish an evidence-based, cost-effective regimen that effectively prevents rejection and minimizes side effects.

Corticosteroid eye drops are the mainstay of ocular immunomodulatory therapy. Their main side effect is a steroid-induced increase in intraocular pressure (IOP). It manifests in about one-fourth of patients within the first year after surgery and can lead to irreversible optic nerve damage and vision loss. Patients with IOP elevation require additional medications and hospital visits resulting in reduced quality of life and increased costs. The optimal dosing regimen in the first year after DMEK and whether patients may safely stop steroids after one year remains unknown. As a result, protocols in the Netherlands vary considerably from surgeon to surgeon. Patients are potentially over-treated in the short and long-term, resulting in undue burden for the patient and increased costs. Consequently, the Dutch Ophthalmology Society (NOG) identified the optimal short- and long-term immunosuppressive protocol for corneal transplantation as one of its Top 10 knowledge gaps, underscoring relevance for clinical practice. With this work, the investigators expect to address this knowledge gap to the benefit of our patients and society.

Objective:

The OPTIMISE study aims to establish an evidence-based, cost-effective regimen that effectively prevents rejection and minimizes side effects. The hypothesis of this study is that Fluorometholone 0.1% in the first year and discontinuing medication in the second year is a cost-effective treatment strategy after DMEK.

Study design:

The design of this study is a randomized, controlled multicentre trial with a duration of 24 months.

Study population:

The study population will consist of 342 patients aged 21 years or older undergoing DMEK surgery in one eye.

Intervention:

All patients will receive Descemet's Membrane Endothelial Keratoplasty. Following this procedure, patients will be randomized into the following post-operative regime in two stages:

STEP-I (Year 1):

Control group: DMS 0.1% 6 times a day for 1 month tapered off to once daily within 6 months and then once a day for 6 months.

Intervention group: DMS 0.1% 6 times a day for 1 month followed by FML 0.1% 4 times a day for two months tapered off to once daily within four months and then once a day for 6 months.

STEP-II (Year 2):

Control Group: Half the patients in each study arm will use FML 0.1% daily. Intervention Group: Half the patients in each study arm will discontinue steroids.

Main study parameters/endpoints:

Primary outcomes:

Step-I: IOP elevation compared to baseline Step-II: Endothelial cell loss (ECL) in the second year

Secondary outcomes are:

* Rejection free graft survival.
* Patient reported outcome measures.
* Incremental cost-effectiveness ratios, including a short term trial-based economic evaluation (TBEE) and a life-long model-based economic evaluation (MBEE)
* Structural outcomes including corneal, central macular and retinal nerve fibre layer thicknesses, and optic nerve head imaging.

ELIGIBILITY:
Inclusion Criteria:

- Patients aged 21 years or older registered on the NOTR as candidates for DMEK corneal transplantation

Exclusion Criteria:

* Inability to complete follow up or comply with study procedures
* The participant is vulnerable
* Previous corneal graft in the study eye
* Known sensitivity or contraindication to the ingredients in the study medications
* History of uveitis
* History of any herpes simplex infection
* Human Leukocyte Antigen (HLA) typed allograft
* Pregnancy (current and planned) or lactation
* Use of other local or systemic immunosuppressive drugs

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Estimated)
Dates: Start 2024-07-29 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Difference of intraocular pressure elevation between the two arms | Year 1
Difference of endothelial cell loss (ECL) in the second year | Year 2

SECONDARY OUTCOMES:
Difference of rejection free graft survival between arms | 1-2 years
Differences of patient reported outcome measures between groups | 1-2 years
Differences of incremental cost-effectiveness ratios, including a short term trial-based economic evaluation (TBEE) and a life-long model-based economic evaluation (MBEE) | 1-2 years

CONTACTS AND LOCATIONS:
Locations (8):
- Netherlands (8):
  - Gelre Ziekenhuizen, Apeldoorn, Gelderland
  - Radboud Universitair Medisch Centrum, Nijmegen, Gelderland
  - Maastricht Universitair Medisch Centrum+, Maastricht, Limburg
  - Amsterdam Universitair Medisch Centrum, Amsterdam, North Holland
  - Deventer Ziekenhuis, Deventer, Overijssel
  - Universitair Medisch Centrum Groningen, Groningen, Provincie Groningen
  - Leiden Universitair Medisch Centrum, Leiden, South Holland
  - Universitair Medisch Centrum Utrecht, Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No